CLINICAL TRIAL: NCT05070975
Title: Phenotype Severity of RSV-infections in Twins During the First Year of Life
Brief Title: Severity of RSV Infections in Twins
Acronym: TwinSeVeRS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0634
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: RSV Infection; Bronchiolitis
Keywords: RSV infections in twins; Bronchiolitis; very-severe-LRTI; severe-LRTI; LRTI; upper respiratory tract infection; RSV infection; Human; infant
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Twins: Twins identified from the birth cohort (Hospices Civils de Lyon) with at least one twin hospitalized for an acute RSV-infection
  Interventions: Other: Epidemiology

INTERVENTIONS:
Other: Epidemiology — Assessment of the discrepancy of clinical severity of RSV-infections between twin infants.

SUMMARY:
Respiratory syncytial virus (RSV) infection is the most common cause of severe lower respiratory tract infection (LRTI) in the pediatric population worldwide. Age at the time of infection, prematurity, multiparity, exposure to smoke and the level of passive immunity transmitted at birth are the main risk factors for lower respiratory infection associated with RSV. Other factors, including the innate immune response, respiratory microbiota, and intra-host viral heterogeneity, may also affect outcomes but are not fully considered in RSV infection. Exploring the impact of these factors is difficult due to the heterogeneity of the population which makes statistical adjustment difficult. Thus, twin models are useful in understanding the impact of the host on the environment, as twins often share similar exposure to infection and many risk factors, but not all are ie different prenatal and postnatal conditions, differential transfer of maternal antibodies and the genetic makeup of heterozygotes.

ELIGIBILITY:
Inclusion Criteria:

* Twins born at Hospices Civils de Lyon in the years 2012 to 2020
* At least one twin hospitalized with positive RSV-PCR during the first year of life

Exclusion Criteria:

* Major differential underlying disease between twins
* Death of a twin before the RSV epidemic period of the first year of life
* Nosocomial infection
* Lack of understanding of the study or questionnaire by parents
* Lack of parental consent

Max Age: 354 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Twins identified from the birth cohort (Hospices Civils de Lyon) with at least one twin hospitalized for an acute RSV-infection
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Percentage of discordant twin pairs in severity of Respiratory Syncytial Virus infections. | 1 day
  The primary outcome measure is the percentage of discordant twin pairs of at least one severity level on the WHO (World Health Organization) scale.
  The discrepancy in the level of severity is obtained by retrospective analysis of the data from the medical file.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme-Mère-Enfant des Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No